CLINICAL TRIAL: NCT00761215
Title: A Phase 2 Multi-Center, Randomized, Double-Blind, Non-Controlled Study Comparing the Safety, Tolerance, and Efficacy of TR-701 in Patients With Complicated Skin and Skin Structure Infections
Brief Title: Phase 2 Study of TR-701 in Patients With Complicated Skin and Skin Structure Infections
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Trius Therapeutics LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1986-007; TR701-104 (Other: TriusRX Unique ID)
Record Dates: First submitted 2008-09-25; First posted 2008-09-29 (Estimated); Results first posted 2014-08-07 (Estimated); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Skin Diseases, Infectious; Skin Diseases, Bacterial
Keywords: Skin; Infection; Complicated Skin and Skin Structure Infection
MeSH Terms: conditions — Skin Diseases, Infectious; Skin Diseases, Bacterial; Infections | interventions — tedizolid phosphate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- TR-701 200 mg (Experimental)
  Interventions: Drug: TR-701 200 mg
- TR-701 300 mg (Experimental)
  Interventions: Drug: TR-701 300 mg
- TR-701 400 mg (Experimental)
  Interventions: Drug: TR-701 400 mg

INTERVENTIONS:
Drug: TR-701 200 mg — oral TR-701 200 mg for 5 to 7 days
  Arms: TR-701 200 mg
Drug: TR-701 300 mg — oral TR-701 300 mg for 5 to 7 days
  Arms: TR-701 300 mg
Drug: TR-701 400 mg — TR-701 400 mg for 5 to 7 days
  Arms: TR-701 400 mg

SUMMARY:
The purpose of the study is to determine the oral dosage of TR-701 to be used in Phase III studies in patients with complicated skin and skin structure infections.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with complicated skin and skin structure infection with at least 2 signs and symptoms
* Suspected or confirmed infection due to a gram-positive organism

Exclusion Criteria:

* Complicated skin and skin structure infection due to gram-negative organisms
* Complicated skin and skin structure infections requiring more than 7 days of therapy
* Uncontrolled diabetes
* Chronic systemic immunosuppressive therapy
* AIDS with CD4 count < 200 cells/mm3
* Uncontrolled hypertension
* Mild moderate or severe renal failure
* Severe hepatic disease
* Neutropenia
* Use of antidepressants such as SSRIs or MAOIs for 14 days before first dose of study drug
* Women who are pregnant or nursing

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2008-09-17 (Actual); Primary Completion 2009-02-24 (Actual); Study Completion 2009-02-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Prokocimer, MD, Study Chair — Trius
Locations (12):
- United States (12):
  - Trius Study Site #011, Dothan, Alabama
  - Trius Study site #001, Chula Vista, California
  - Trius Study Site #009, Long Beach, California
  - Trius Study site #002, Oceanside, California
  - Trius Study site #010, Pasadena, California
  - Trius Study site 007, San Francisco, California
  - Trius Study site 003, San Jose, California
  - Trius Study site 004, Columbus, Georgia
  - Trius Study site #006, Ludowici, Georgia
  - Trius Study site #005, Savannah, Georgia
  - Trius Study site #012, Springfield, Illinois
  - Trius study sie #008, Detroit, Michigan

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Prokocimer P, Bien P, Deanda C, Pillar CM, Bartizal K. In vitro activity and microbiological efficacy of tedizolid (TR-700) against Gram-positive clinical isolates from a phase 2 study of oral tedizolid phosphate (TR-701) in patients with complicated skin and skin structure infections. Antimicrob Agents Chemother. 2012 Sep;56(9):4608-13. doi: 10.1128/AAC.00458-12. Epub 2012 Jun 11. PMID 22687509

RESULTS

PARTICIPANT FLOW:
Groups:
- TR-701 200 mg: Oral TR-701 200 mg once daily for 5 to 7 days
- TR-701 300 mg: Oral TR-701 300 mg once daily for 5 to 7 days
- TR-701 400 mg: Oral TR-701 400 mg once daily for 5 to 7 days
Period: Overall Study
Arm/Group | TR-701 200 mg | TR-701 300 mg | TR-701 400 mg
Started | 64 | 64 | 64
Completed | 55 | 60 | 56
Not Completed | 9 | 4 | 8
Not completed — Randomized but didn't receive drug | 1 | 1 | 2
Not completed — Lost to Follow-up | 6 | 3 | 6
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Bacteremia | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants who received study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | TR-701 200 mg | TR-701 300 mg | TR-701 400 mg | Total
Number analyzed (Participants) | 63 | 63 | 62 | 188
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.3 (12.1) | 36.0 (12.4) | 35.8 (12.0) | 36.4 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 24 | 22 | 66
  Male | 43 | 39 | 40 | 122

OUTCOME MEASURES:

1. Primary Outcome: Clinical Response Rate at Test of Cure in the Clinically Evaluable Analysis Set
Description: Clinical response was defined as resolution or improvement of signs and symptoms of the complicated skin and skin structure infection so that no further antibiotic therapy was required.
Time Frame: 7 to 14 days after the last dose of study drug
Population: The Clinically Evaluable analysis set includes data from all participants who had a diagnosis of cSSSI, received minimal study therapy, completed an assessment, and had no confounding events or factors.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- TR-701 400 mg: Oral TR-701 400 mg for 5 to 7 days
Arm/Group | TR-701 200 mg | TR-701 300 mg | TR-701 400 mg
Number analyzed (Participants) | 56 | 54 | 54
Percentage of participants | 98.2 [90.4 to 100] | 94.4 [84.6 to 98.8] | 94.4 [84.6 to 98.8]

2. Primary Outcome: Clinical Response Rate at Test of Cure in the Clinical Modified Intent to Treat Analysis Set
Description: as for outcome 1
Time Frame: 7-14 days after last dose of study drug
Population: The clinically modified intent to treat analysis set includes data from all participants who received study drug and had a diagnosis of complicated skin and skin structure infection.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | TR-701 200 mg | TR-701 300 mg | TR-701 400 mg
Number analyzed (Participants) | 63 | 63 | 62
Percentage of participants | 88.9 [78.4 to 95.4] | 88.9 [78.4 to 95.4] | 85.5 [74.2 to 93.1]

3. Secondary Outcome: Response Rate at End of Therapy
Description: as for outcome 1
Time Frame: last day of study treatment
Population: The clinical modified intent to treat analysis set includes data from all participants who received study drug and had a diagnosis of complicated skin and skin structure infection
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | TR-701 200 mg | TR-701 300 mg | TR-701 400 mg
Number analyzed (Participants) | 63 | 63 | 62
Percentage of participants | 93.7 [84.5 to 98.2] | 90.5 [80.4 to 96.4] | 91.9 [82.2 to 97.3]

4. Secondary Outcome: Microbiological Response Rate at Test of Cure in the Microbiologically Evaluable Analysis Set
Description: Satisfactory microbiological outcomes are eradication and presumed eradication
Time Frame: 7-14 days after last dose of study drug
Population: The microbiologically evaluable analysis set includes all participants who received study drug, had a diagnosis of complicated skin and skin structure infection, completed an assessment, had no confounding events or factors, and had a baseline Gram-positive bacterial pathogen.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | TR-701 200 mg | TR-701 300 mg | TR-701 400 mg
Number analyzed (Participants) | 43 | 44 | 46
Percentage of participants | 100 [91.8 to 100] | 93.2 [81.3 to 98.6] | 100 [92.3 to 100.0]

5. Secondary Outcome: Clinical Outcome at the Late Follow-up Visit in the Clinical Modified Intent to Treat Analysis Set
Description: Persistent clinical cure was defined as continuing favorable response.
Time Frame: 21 to 28 days after the last study drug
Population: The clinical modified intent to treat analysis set includes data from all participants who received study drug and had a diagnosis of complicated skin and skin structure infection. Microbiological samples not available from all participants.
Measure: Number; unit: Percentage of Participants
Arm/Group | TR-701 200 mg | TR-701 300 mg | TR-701 400 mg
Number analyzed (Participants) | 56 | 56 | 53
Percentage of Participants | 96.4 | 98.2 | 98.1

6. Secondary Outcome: To Evaluate the Safety Profile of Tedizolid Phosphate
Time Frame: Multiple
Reporting Status: Not Posted

7. Secondary Outcome: Population PK
Time Frame: Multiple
Reporting Status: Not Posted

8. Secondary Outcome: Microbiological Recurrence at Late Follow-up in Clinical Modified Intent to Treat Analysis Set
Time Frame: 21-28 days after last study drug
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | TR-701 200 mg | TR-701 300 mg | TR-701 400 mg
Number analyzed (Participants) | 56 | 56 | 53
Percentage of participants | 0 [0 to 6.4] | 0 [0 to 6.4] | 0 [0 to 6.7]

ADVERSE EVENTS:
Time Frame: Adverse events were to be collected after informed consent through last visit (up to 36 days).
Arm/Group | TR-701 200 mg | TR-701 300 mg | TR-701 400 mg
Serious Adverse Events (participants affected / at risk) | 2/63 | 1/63 | 2/62
Other Adverse Events (participants affected / at risk) | 40/63 | 44/63 | 43/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TR-701 200 mg (N=63) | TR-701 300 mg (N=63) | TR-701 400 mg (N=62)
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 1
Abcess (Infections and infestations) | 1 | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TR-701 200 mg (N=63) | TR-701 300 mg (N=63) | TR-701 400 mg (N=62)
Tachycardia (Cardiac disorders) | 2 | 1 | 1
Diarrhea (Gastrointestinal disorders) | 7 | 3 | 6
Dry mouth (Gastrointestinal disorders) | 0 | 2 | 2
Nausea (Gastrointestinal disorders) | 10 | 12 | 13
Vomiting (Gastrointestinal disorders) | 7 | 6 | 6
Fatigue (General disorders) | 3 | 1 | 1
Pain (General disorders) | 2 | 2 | 2
Abscess (Infections and infestations) | 5 | 8 | 7
Skin infection (Infections and infestations) | 4 | 2 | 2
Blood pressure increased (Investigations) | 1 | 4 | 2
Decreased appetite (Metabolism and nutrition disorders) | 1 | 2 | 2
Dizziness (Nervous system disorders) | 4 | 1 | 0
Headache (Nervous system disorders) | 5 | 10 | 6
Insomnia (Psychiatric disorders) | 1 | 4 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 2 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 2 | 2
Skin lesion (Skin and subcutaneous tissue disorders) | 4 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor intends to pursue publication of the results of the study in cooperation with a lead Investigator, subject to the terms and conditions of the clinical trial agreement between Sponsor and Investigators. Sponsor approval is required for publication of any data subsets. Final authorship will be determined by contributions to study design, enrollment, data analysis, and/or interpretation of the results.